CLINICAL TRIAL: NCT07299279
Title: Movement Improves Brain Health and Cognition in Parkinson's Disease
Acronym: MOVE-BRAIN-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7536
Record Dates: First submitted 2025-05-14; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (EG) (Experimental): The EG will be prescribed aerobic exercise for >_ 75 minutes/week of vigorous aerobic exercise (60%-85% of HR MAX) or >_150 minutes/week of moderate aerobic exercise (40%-60% of HR MAX) in at least two weekly sessions, for 12 months.
  Interventions: Behavioral: Aerobic exercise for >_75 minutes/week of vigorous aerobic exercise or >_ 150 minutes/week of moderate aerobic exercise in at least two weekly sessions, for 12 m
- Sedentary group (SG) (No Intervention): The SG will be told to continue their routine daily activities and will be followed up regularly at the outpatient clinic.

INTERVENTIONS:
Behavioral: Aerobic exercise for >_75 minutes/week of vigorous aerobic exercise or >_ 150 minutes/week of moderate aerobic exercise in at least two weekly sessions, for 12 m — Participants will use a commercially available wearable device with a heart rate monitor to prove adherence to the program and record the intensity of all exercise sessions.
  Arms: Exercise group (EG)

SUMMARY:
Cognitive impairment is an acknowledged feature of Parkinson's disease (PD) and often coexists with the classic motor symptoms since their onset. Cognitive symptoms of PD can be differentiated from other neurodegenerative diseases by the affected domains: typically, the executive functions are primarily affected, to a greater extent than the mnesic ones. PD-MCI is of utmost clinical relevance, as it impacts the patients' quality of life and as the major predictor for conversion to PDD. To date, there are no routinely recommended interventions to address MCI in PD and prevent it from evolving into dementia. Recent evidence supports the benefit of aerobic exercise on motor symptoms of PD and its possible disease-modifying role, through functional and structural brain changes. Less is known about the impact of aerobic exercise on cognition in the PD population. In the last decade, studies have proven aerobic exercise as a promising strategy to alter the trajectory of cognitive decline in subjects with cognitive impairment and in elderly people. In particular, executive functions were ameliorated by exercise intervention to a greater extent. A recent preclinical study also demonstrated a reduced spread of toxic alpha-synuclein (a-syn) species to vulnerable brain areas, along with the restoration of the striatal synaptic plasticity. Nonetheless, the feasibility and efficacy of an unsupervised monitored exercise program on cognition for PD-MCI subjects has not been explored yet. In this project, we will test the hypothesis that extensive homebased exercise may improve cognition in MCI-PD through a reduction of neuroinflammation and a-syn spreading via the activation of BDNF-related pathways. Motor, non-motor and cognitive evaluations, associated with measures of a-syn species, inflammation-related molecules and neurofilaments light chain in blood samples will be performed in a multicenter cohort, before and after the prescription of moderate/vigorous aerobic home-based exercise for 12 months and in a sedentary control population. Adherence to the protocol will also be evaluated. This will shed light on the impact of physical activity prescription in the care of people with PD, addressing one of the most unmet needs in PD, since no disease-modifying treatments are available for cognitive deficits to date.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 30 and 80 years, with a clinical diagnosis of Parkinson's disease (PD) according to the Movement Disorder Society (MDS) diagnostic criteria and a Hoehn & Yahr (H&Y) stage between 1 and 3, as well as a diagnosis of mild cognitive impairment (MCI) according to MDS-PD-MCI level II criteria, will be consecutively enrolled during routine clinical practice at the hospitals of the Principal Investigator (PI) and Partner
2. The inclusion criteria for the study's physical activity intervention are based on the guidelines of the American College of Sports Medicine. To be eligible for the study, potential participants must not engage in more than 120 minutes/week of moderate-intensity exercise or more than 60 minutes/week of vigorous-intensity exercise. Enrolled patients must be able to provide informed consent to participate in the study.

Exclusion Criteria:

* Pregnant patients, patients with medical conditions that prevent vigorous physical exercise, those with oncological or autoimmune comorbidities, or those taking immunomodulatory or anti-inflammatory medications will be excluded from the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Motor performance | From enrollment (time 0) to the end of exercise (after 12 months)
  · Unified Parkinson's Disease Rating Scale - MDS (MDS-UPDRS) to evaluate various aspects of PD, including non-motor and motor experiences of daily living and motor complications (0-272, the higher, the worse)
non motor assessment | From enrollment (time 0) to the end of exercise (after 12 months)
  · MDS - Non-Motor Symptoms Rating Scale (MDS-NMS) which measures the severity and frequency of non-motor symptoms (0-360, the higher, the worse)
disease stage | From enrollment (time 0) to the end of exercise (after 12 months)
  · Hoehn and Yahr stage (H&Y), to assess disease stage (1-4, the higher the worse)
Cognitive evaluation | From enrollment (time 0) to the end of exercise (after 12 months)
  . Montreal Cognitive assessment (0-30, the lower the worse)

SECONDARY OUTCOMES:
Biochemical analysis of biomarkers | From enrollment (time 0) to the end of exercise (after 12 months)
  Studying changes in biomarkers of inflammation and neurodegeneration in people with Parkinson's disease following a home exercise program (serum levels of IL1B, IL4, IL5, IL6, IL10, IL17, IFN-gamma, TNF-alpha, total alpha synuclein)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Calabresi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Rome, Italy